CLINICAL TRIAL: NCT05512325
Title: Study on Gene Evolution and Anti-VEGF Treatment Response of Different Subtypes of Glioma Based on ctDNA
Brief Title: Study on Gene Evolution in Glioma Under Stress Therapy
Status: Not yet recruiting | Type: Observational
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HenanPPH-GRS
Record Dates: First submitted 2022-08-21; First posted 2022-08-23 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-08

CONDITIONS: Genetic Change
Keywords: gene evolution, ctDNA, molecular response, Bevacizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — A small amount of TISF was harvested from the implanted reservoir(Intra-operative retention) during postoperative progression of 20 glioma patients under stress therapy. At the same time, blood samples (5ml) for germline DNA control were also acquired. Fresh tumor tissues were obtained for comparing evolution analysis with TISF ctDNA under bevacizumab treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gene evolution of glioma in vivo: Group A: gene evolution with relapsed. From the first day after the operation, the ctDNA was extracted from TISF before concurrent chemoradiotherapy as the baseline, and then the ctDNA was detected again after concurrent chemoradiotherapy. For the third time, ctDNA was detected in intensive chemotherapy with temozolomide. The image showed that the tumor progress was detected for the fourth time, and the ctDNA was detected for the fifth time when the tumor recurred. Patients with glioma were routinely treated with temozolomide chemotherapy from the 4th week after operation, for 5 days continuously, once every 4 weeks, with a single dose as follows: Single dose = BSA (body surface area) * 150mg/m2/day BSA(Body Surface Area)=[weight (kg)* height (cm)/3600]2,
- Gene evolution and molecular response under Bevacizumab treatment: After the recurrence, temozolomide combined with bevacizumab was used for chemotherapy, After bevacizumab was applied after six week , ctDNA is tested every six weeks. temozolomide combined with bevacizumab (600mg) in the course of tumor progression once a month.
  Interventions: Drug: Gene evolution and molecular response under Bevacizumab treatment

INTERVENTIONS:
Drug: Gene evolution and molecular response under Bevacizumab treatment — Patients with glioma were routinely treated with temozolomide chemotherapy from the 4th week after operation, for 5 days continuously, once every 4 weeks, with a single dose as follows: Single dose = BSA (body surface area) * 150mg/m2/day BSA(Body Surface Area)=[weight (kg)* height (cm)/3600]2, According to the molecular pathological grade (WHO CNS5 grade), it is decided whether to combine radiotherapy (GBM combined with radiotherapy) and temozolomide combined with bevacizumab (600mg) in the course of tumor progression, Recording image changes
  Groups: Gene evolution and molecular response under Bevacizumab treatment

SUMMARY:
Little is known about the evolution of genetic and epigenetic changes that occur in the progression of glioma. We inferred the evolution trajectories of matched pairs of primary tumors and progression tumor in situ fluid (TISF) based on deep whole-genome-sequencing data (ctDNA). A monocentric, Gene grouping controlled trial design was used to select patients. and to compare gene evolution of different subtypes of glioma under therapy. To predict the molecular reaction of bevacizumab treatment, clarify the mechanism of drug resistance of bevacizumab treatment.

DETAILED DESCRIPTION:
Patient: Adult glioma, pathological diagnosis combined with molecular diagnosis (i.e. IDH- mutant glioma, IDH- mutant glioma with 1p/19q- co-deletion, glioblastoma). The patients were divided into three groups: group A (IDH mutant glioma), group B (IDH mutant with 1p/19q co-deletion oligodendroglioma ) and group C (IDH wild glioblastoma). From the first day after surgery, the ctDNA was extracted with TISF before concurrent chemoradiotherapy as the baseline, and the ctDNA was detected again after concurrent chemoradiotherapy. For the third time, ctDNA was detected in temozolomide intensive chemotherapy. ctDNA was detected for the fourth time when the image showed tumor progression. After the progress, temozolomide combined with bevacizumab was used for chemotherapy. ctDNA was detected 6 weeks after the application of bevacizumab, and ctDNA was re-measured every 6 weeks during the treatment of bevacizumab. At the same time, imaging examination was performed to determine the tumor progress. Check and record adverse events and drug use in detail, and evaluate the compliance of subjects; After TISF tissue extraction, the retained blood samples were sent to simcere Company and Beijing Genetron Health Technology Co. Ltd for ctDNA quantification and detection. To study the differences of gene evolution of different subtypes of glioma under pressure therapy, to clarify the differences of molecular responses of different subtypes of glioma to bevacizumab, and to evaluate the therapeutic effect and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years, both male and female (including 18 and 75 years old) glioma;
* Willing to accept treatment and sign informed consent.

Exclusion Criteria:

* Participants with other infection disease or immunodeficiency disease;
* other central infectious diseases;
* malignant tumor of non-nervous system;
* drug abuse;
* severe psychiatric disease;
* uncontrolled diabetes;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age 18 to 75 years, both male and female (including 18 and 75 years old) glioma; Willing to accept treatment and sign informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-17 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Different subtypes of glioma have different therapeutic responses to bevacizumab | 96 weeks
  We evaluated the efficacy of bevacizumab on different subtypes of glioma at recurrence according to delta-VAF and Ratio combined with imaging.The mean change in VAF (delta-VAF) was calculated per patient as the sum of the ontreatmentVAF minus the pretreatment VAF for each detected SNV or indel divided by the number of detected SNVs or indels, we found that the "molecular responce" model could generally be represented in simpler terms through a ratio of ontreatment VAF to pretreatment VAF
the molecular mechanism of bevacizumab resistance in vivo. | 144 weeks
  We compared and analyzed the genes before and after bevacizumab treatment according to the gene evolution of ctDNA.To clarify the molecular mechanism of bevacizumab resistance.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu G, Bu C, Guo G, Zhang Z, Sheng Z, Deng K, Wu S, Xu S, Bu Y, Gao Y, Wang M, Liu G, Kong L, Li T, Li M, Bu X. Molecular and clonal evolution in vivo reveal a common pathway of distant relapse gliomas. iScience. 2023 Aug 2;26(9):107528. doi: 10.1016/j.isci.2023.107528. eCollection 2023 Sep 15. PMID 37649695
- [Derived] Liu G, Bu C, Guo G, Zhang Z, Sheng Z, Deng K, Wu S, Xu S, Bu Y, Gao Y, Wang M, Liu G, Kong L, Li T, Li M, Bu X. Genomic alterations of oligodendrogliomas at distant recurrence. Cancer Med. 2023 Aug;12(16):17171-17183. doi: 10.1002/cam4.6327. Epub 2023 Aug 2. PMID 37533228